CLINICAL TRIAL: NCT06203106
Title: NYSCF Scientific Discovery Biobank
Status: Recruiting | Type: Observational
Sponsor: New York Stem Cell Foundation Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 10-010
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: ALS; Amyotrophic Lateral Sclerosis; Alzheimer Disease; Alzheimer Disease, Early Onset; Alzheimer Disease, Late Onset; Batten Disease; Corticobasal Degeneration; Dementia; Frontotemporal Dementia; Huntington Disease; Lewy Body Disease; Multiple Sclerosis; Multiple System Atrophy; Parkinson Disease; Parkinson's Disease and Parkinsonism; Progressive Supranuclear Palsy; INAD; Diabetes; Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Macular Degeneration; Ovarian Cancer; Cervical Cancer; Uterine Cancer; Vaginal Cancer; Vulvar Cancer; PTSD; Post Traumatic Stress Disorder
Keywords: ALS; Amyotrophic Lateral Sclerosis; Alzheimer Disease; Batten Disease; Corticobasal Degeneration; Dementia; Frontotemporal Dementia; Huntington Disease; Lewy Body Disease; Multiple Sclerosis; Multiple System Atrophy; Parkinson Disease; Parkinsonism; Progressive Supranuclear Palsy; INAD; Diabetes; Diabetes Type 1; Diabetes Type 2; Macular Degeneration; Women's Reproductive Cancer; Ovarian Cancer; Cervical Cancer; Uterine Cancer; Vaginal Cancer; Vulvar Cancer; PTSD; Post Traumatic Stress Disorder
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Alzheimer Disease; Neuronal Ceroid-Lipofuscinoses; Corticobasal Degeneration; Dementia; Frontotemporal Dementia; Huntington Disease; Lewy Body Disease; Multiple Sclerosis; Multiple System Atrophy; Parkinson Disease; Parkinsonian Disorders; Supranuclear Palsy, Progressive; Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Macular Degeneration; Ovarian Neoplasms; Uterine Cervical Neoplasms; Uterine Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin biopsy (2-3mm) and/or blood (up to 50 mL); saliva; excess/leftover biospecimens that were (or will be) collected for other purposes (e.g., medical procedure)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Affected Subjects: Subjects in this group will have a diagnosis and/or medical history of a condition, disease, genetic background, or trait of interest.
  Interventions: Other: Biological Sample Collection
- Healthy Control: Subjects in this group will serve as healthy controls.
  Interventions: Other: Biological Sample Collection

INTERVENTIONS:
Other: Biological Sample Collection — Skin biopsy (2-3mm) and/or blood (up to 50 mL); saliva; excess/ leftover biospecimens that were (or will be) collected for other purposes (e.g., medical procedure).

SUMMARY:
The New York Stem Cell Foundation (NYSCF) Research Institute is performing this research to accelerate diverse disease research using cells from the body (such as skin or blood cells) to make stem cells and other types of cells, conduct research on the samples, perform genetic testing, and store the samples for future use.

Through this research, researchers hope to identify future treatments or even cures for the major diseases of our time.

DETAILED DESCRIPTION:
Researchers at the New York Stem Cell Foundation (NYSCF) Research Institute study diverse diseases, conditions, and traits by creating stem cells from biological samples. These "pluripotent" stem cells can become any cell in the human body, including cells that may be difficult, invasive, or impossible to obtain directly.

Additionally, researchers perform genetic testing to learn more about DNA, a material in most cells that contains instructions for the body's development and functions (such as traits like eye color and risk of certain diseases). A piece of DNA that determines the specific role of a cell is called a "gene." If the instructions in a gene are abnormal, this can lead to disease.

Participation in the study involves: (1) completion of health questionnaires, (2) providing a skin and/or blood sample from which stem cells may be created, (3) collection of a saliva sample for genetic analysis, and (4) possible future followup to provide additional information or learn about other research studies.

This study is not a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 days or older.
* Diagnosis and/or medical history of a condition, disease, genetic background, or trait of interest or healthy control.
* Adults with decisional capacity must provide written informed consent unless physical limitations preclude signing.
* Adults without decisional capacity to consent must a have diagnosis of Amyotrophic Lateral Sclerosis (ALS), Alzheimer's Disease and Related Dementias (AD/ADRD); Batten Disease, Corticobasal Degeneration (CBD), Dementia, Frontotemporal Dementia (FTD), Huntington Disease, Lewy Body Disease, Multiple Sclerosis, Multiple System Atrophy, Parkinson's Disease (PD), Parkinsonism, and/or Progressive Supranuclear Palsy, and must provide assent; a legally authorized representative (LAR) must also provide written informed consent.
* Minors undergoing skin collection for research purposes must have a condition, disease, genetic background, or trait of interest and parental/guardian consent.
* Minors undergoing blood, and/or saliva collection for research purposes may have a condition, disease, genetic background, or trait of interest or serve as a healthy control and must have an available parent/guardian to provide consent.
* Minors transferring biological samples and associated data from a procedure outside of the research may have a condition, disease, genetic background, or trait of interest or serve as a healthy control and must have an available parent/guardian to provide consent.

Exclusion Criteria:

* Wards of the state.
* For prospective skin samples: history of keloid formation, coagulation disorder, or allergy to the anesthetic.
* For prospective blood samples: history of coagulation disorder.
* For all prospective sample collections: 1) Subjects who refuse to adhere to NYSCF's and/or a collection site's safety protocol(s) will be excluded; 2) Subjects with an AIDS diagnosis and CD4 count of less than 200 cells per microliter (mcL) of blood will be excluded due to increased risk of infection.

Min Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a diagnosis of one or more of the listed conditions. Individuals without a condition to serve as healthy controls (a comparison group for those with conditions).
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2045-11-10 (Estimated); Study Completion 2045-11-10 (Estimated)

PRIMARY OUTCOMES:
Biobank | Baseline
  Establishment of a diverse repository of biological samples, stem cell lines, derivatives, and associated information to support investigations into the biology, etiology, manifestations, progression, risk factors, genetic underpinnings, and treatment of diseases, conditions, and traits.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Andres-Martin, PhD, Principal Investigator — New York Stem Cell Foundation Research Institute
Locations (1):
- New York Stem Cell Foundation Research Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No